CLINICAL TRIAL: NCT04093245
Title: Supporting the Creation of a LEARNing INteGrated Health System to Mobilize Context-adapted Knowledge With a Wiki Platform to Improve the Transitions of Frail Seniors From From Hospitals and Emergency Departments to the cOMmunity: Phase II
Brief Title: The LEARNING WISDOM Phase II Scale up Project
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Patrick Archambault, Associate Professor, Laval University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: Learning Wisdom 2018-462
Record Dates: First submitted 2019-09-09; First posted 2019-09-17 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Transition; Emergencies; Health Care Utilization; Frailty
Keywords: Emergency Department; Care Transition; Elderly Frailty
MeSH Terms: conditions — Emergencies; Patient Acceptance of Health Care; Frailty | interventions — Lead

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase I-A (Local project set-up) (No Intervention): An executive committee will oversee the entire project. This committee, led by the nominated PI and Director of Nursing, will meet every 4 weeks during this four-year project. The team may include, depending on the hospital site: an administrator, the ED Director, the ED Head nurse, a community and/or hospital-based geriatric nurse specialist, an ED physician, a hospitalist, a geriatrician, a family physician, a home care nurse/coordinator, an inpatient unit manager, the research coordinator, and a local patient/caregiver. Each local team will be responsible for selecting and implementing the ACE intervention(s) best suiting their milieu, and will include locally identified champions to lead the local implementation.
- Phase I-B (Implementation): (Experimental): The investigators will implement the context-adapted ACE program with the support of administrators and local implementation teams who will have the responsibility to roll out the different elements of the intervention within their respective hospitals. It may include a series of systematic pre-discharge, post-discharge and across transitions period interventions for eligible patients: 1) a GEM nurse to support patients during the post-discharge transition period, 2) pre- and post-hospitalization medication list reconciliation, 3) systematic discharge summaries given to patients and/or caregiver, and sent to their family physician, 4) a planned follow-up appointment with their family physician, 5) a systematic follow-up phone call, 6) access to wiki-based patient-oriented KT tools, 7) access to a community-based telemonitoring service.
  Interventions: Behavioral: GEM nurse; Behavioral: pre- and post-hospitalization medication list reconciliation; Behavioral: systematic discharge summaries; Behavioral: medical follow-up appointment; Behavioral: follow-up phone call; Other: Wiki-based Knowledge tools; Other: Telemonitoring service
- Phase IC (Study description) (Experimental): Results from each center will be analysed over time. Guided by previous work in healthcare governance, the investigators will analyze the impact of the sequential interventions within the context of a major health reform in Quebec aiming at implementing an integrated health system and within the PI program's overall goal of creating a Learning Health System. This will be accomplished by conducting a comparative case study across the four study sites to compare the barriers, facilitators and local solutions implemented to gain a better understanding about how the ACE program could eventually be scaled up elsewhere.
  Interventions: Behavioral: GEM nurse; Behavioral: pre- and post-hospitalization medication list reconciliation; Behavioral: systematic discharge summaries; Behavioral: medical follow-up appointment; Behavioral: follow-up phone call; Other: Wiki-based Knowledge tools; Other: Telemonitoring service

INTERVENTIONS:
Behavioral: GEM nurse — hospital-based geriatric emergency nurse (GEM nurse) specialist to support patients during the post-discharge transition period
  Arms: Phase I-B (Implementation):; Phase IC (Study description)
Behavioral: pre- and post-hospitalization medication list reconciliation — pre- and post-hospitalization medication list reconciliation for elderly
  Arms: Phase I-B (Implementation):; Phase IC (Study description)
Behavioral: systematic discharge summaries — systematic discharge summaries given to patients and/or caregiver, and sent to their family physician
  Arms: Phase I-B (Implementation):; Phase IC (Study description)
Behavioral: medical follow-up appointment — a planned follow-up appointment with their family physician
  Arms: Phase I-B (Implementation):; Phase IC (Study description)
Behavioral: follow-up phone call — a systematic follow-up phone call for discharged patients
  Arms: Phase I-B (Implementation):; Phase IC (Study description)
Other: Wiki-based Knowledge tools — access to wiki-based patient-oriented KT tools
  Arms: Phase I-B (Implementation):; Phase IC (Study description)
Other: Telemonitoring service — access to a community-based telemonitoring service
  Arms: Phase I-B (Implementation):; Phase IC (Study description)

SUMMARY:
Inspired by the Acute Care for Elders program at Mount Sinai Hospital, this study aims to improve care for elderly patients in four hospitals of Chaudière-Appalaches. Focusing on improving transitions between hospital and the community, this project will help professionals to adapt best practices to local context in transition of care for the elderly.

DETAILED DESCRIPTION:
Background: Elderly patients discharged from hospital currently experience fragmented care, repeated and lengthy emergency department (ED) visits, relapse into their earlier condition, and rapid cognitive and functional decline. The Acute Care for Elders (ACE) program at Mount Sinai Hospital uses innovative strategies such as transition coaches, follow-up calls and patient self-care guides to improve the care transition experiences of the frail elderly patients from hospitals to the community. The ACE program reduced lengths of hospital stay and readmissions for elderly patients, increased patient satisfaction, and saved the healthcare system over $6 million in 2014.

In 2016, the ACE program was implemented at one hospital in the Centre intégré en santé et en services sociaux de Chaudière-Appalaches (CISSS CA), a large integrated healthcare organization in Quebec, with a focus on improving transitions between hospital and the community for the elderly. This project used rapid, iterative user-centered design prototyping and a "Wiki-suite" (a free online database containing evidence-based knowledge tools in all areas of healthcare and an accompanying training course) to engage multiple stakeholders including a patient partner to improve care for elderly patients. Within this one year project, the investigators developed a context-adapted ACE intervention with the support of the Mt. Sinai Hospital, the Canadian Foundation for Healthcare Improvement and the Canadian Frailty Network.

The goal is to scale up the ACE program for elderly care transition to three new hospital sites within the CISSS CA, using the Wiki-suite to allow for further context-adaptation of the program in these new hospitals.

Objectives: 1) Implement a context-adapted ACE program in three hospitals in the CISSS CA and measure its impact on patient, caregiver, clinical and hospital-level outcomes; 2) Identify underlying mechanisms by which the context-adapted ACE program improves care transitions for the elderly; 3) Identify underlying mechanisms by which the Wiki-suite contributes to context-adaptation and local uptake of knowledge tools.

Methods: Objective 1: Staggered implementation of the ACE program across the three CISSS CA sites; interrupted time series to measure the impact on hospital-level outcomes; pre/post cohort study to measure the impact of the new program on patient, caregiver and clinical outcomes. Objectives 2 and 3: Parallel mixed-methods process evaluation study to understand the mechanisms by which the context-adapted ACE program improves care transitions for the elderly and by which the Wiki-suite contributes to adaptation, implementation and scaling up of geriatric knowledge tools.

Expected results: This project will provide much needed evidence on effective Knowledge Translation (KT) strategies to adapt best practices to local context in transition of care for the elderly. It will contribute to adapting geriatric knowledge to local contexts. The knowledge generated through this project will support future scale-up of the ACE program and the wiki methodology to other settings in Canada.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients will be:

* aged ≥ 65 years
* be discharged from the ED
* able to understand and read French
* able to give informed consent

Eligible caregivers will be:

* identified by the patients themselves
* able to understand and read French
* able to give informed consent

Exclusion Criteria:

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2019-01-21 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of 30-day hospital readmission | each month during 4 years (48)
  Composite endpoint at each month 30-day hospital readmission
Change of 30-day ED visit rate | each month during 4 years (48)
  Composite endpoint at each month 30-day ED visit rate

SECONDARY OUTCOMES:
1- change Hospital/ED length of stay - Hospital-level outcome | Each month during 4 years (48)
  Hospital administrative databases (e.g., MedGPS, Logibec, Montreal, Canada) will be used to calculate monthly hospital-level outcomes. Monthly data will then be analyzed to form points in time. Data from the Régie d'assurance maladie du Québec (RAMQ) physician billing database and MedECHO database (containing data on hospitalizations and health professional consultations for all institutions) will also be extracted in addition to databases available at the Institut national d'excellence en santé et services sociaux (INESSS) in order to identify all health services used prior to and after the implementation of the ACE intervention. 1) Hospital/ED length of stay
2- change ED admission rate - Hospital-level outcome | Each month during 4 years (48)
  Hospital administrative databases (e.g., MedGPS, Logibec, Montreal, Canada) will be used to calculate monthly hospital-level outcomes. Monthly data will then be analyzed to form points in time. Data from the Régie d'assurance maladie du Québec (RAMQ) physician billing database and MedECHO database (containing data on hospitalizations and health professional consultations for all institutions) will also be extracted in addition to databases available at the Institut national d'excellence en santé et services sociaux (INESSS) in order to identify all health services used prior to and after the implementation of the ACE intervention. 2) ED admission rate
3- Change Alternate level care occupation rate- Hospital-level outcome | Each month during 4 years (48)
  Hospital administrative databases (e.g., MedGPS, Logibec, Montreal, Canada) will be used to calculate monthly hospital-level outcomes. Monthly data will then be analyzed to form points in time. Data from the Régie d'assurance maladie du Québec (RAMQ) physician billing database and MedECHO database (containing data on hospitalizations and health professional consultations for all institutions) will also be extracted in addition to databases available at the Institut national d'excellence en santé et services sociaux (INESSS) in order to identify all health services used prior to and after the implementation of the ACE intervention. 3) Alternate level care occupation rate
4- Change Rate of patients returning to pre-hospital living situation- Hospital-level outcome | Each month during 4 years (48)
  Hospital administrative databases (e.g., MedGPS, Logibec, Montreal, Canada) will be used to calculate monthly hospital-level outcomes. Monthly data will then be analyzed to form points in time. Data from the Régie d'assurance maladie du Québec (RAMQ) physician billing database and MedECHO database (containing data on hospitalizations and health professional consultations for all institutions) will also be extracted in addition to databases available at the Institut national d'excellence en santé et services sociaux (INESSS) in order to identify all health services used prior to and after the implementation of the ACE intervention. 4) Rate of patients returning to pre-hospital living situation
Clinicians and decision maker outcomes (Qualitative outcome) | each 3 months, during 4 years (12)
  Individual interviews will be performed every 3 months after the beginning of the implementation of the Acute Care for Elders (ACE) program at each hospital among health professionals and decision makers participating in the ACE program. These semi-structured interviews will be based on the National Health Services (NHS) Sustainability Model. This qualitative questionnaire will serve to identify the contextual elements that influenced the successful (or failed) implementation of the (Approche adaptée à la personne âgée) AAPA / ACE program for improving care transitions. These interviews will be conducted by doctoral and/or Master students, guided by experienced qualitative researcher
1- Care Transitions Measure (CTM3) - Patient outcome | 48-72 hours post-discharge for 3-item Care Transitions Measure (CTM3)
  The 3-item Care Transitions Measure (CTM-3) is a 3-item questionnaire measuring the perceived quality of the transition care on a 0-3 scale (0 = fully disagree; 4 = fully agree). Mean of the 3 items are linearized to obtain 0-100 scoring scale.
2- GAI-SC-SF - Patient outcome | within 7 days after post-discharge
  The Geriatric Anxiety Inventory-short form (GAI-SF) has been specifically developed to measure anxiety among seniors and it has good psychometric values. The short version comprises five questions.Each positive item/question = 1. Score range 0 to 5. Anxiety is detected 3 out of 5 and above.
3- Living situation - Patient outcome | 30 days post-discharge
  Living situation will be collected in the medical file when available at 30 days post-discharge.
4- baseline sociodemographic data - Patient outcome | within 7 days after post-discharge
  baseline sociodemographic data (age, sex, race, language, education level, family income will be collected.
Caregiver-level outcomes | 7days patient post-discharge
  The Zarit Burden Interview (ZBI) is one of the most used tools for measuring the burden of caregivers. The brief French version (12 questions) of the scale has good psychometric properties, comparable to the original version.For each question, range answer is : Never=0, Rarely= 1, Sometimes= 2, Quite frequently=3, Nearly always=4. Summation of 12 items 0 to 4 points per item range 0 to 48 as total score. Score between 0-10 = no to mild burden; score between 10-20 = mild to moderate burden; score >20 = high burden.This tool is already used by CISSS-CA staff. Mentioned in Quebec's "Alzheimer's Plan"[89], caregiver burden increases as the disease progresses and is associated with psychological distress and physical health problems. Caregivers are therefore a "risk group" within the health system.
1-Clinical-level process outcome - Proportion of patients assigned a GEM Nurse | Process assessment with a monthly Chart audit for 4 years
  Proportion of patients assigned a GEM Nurse
2-Clinical-level process outcome - Proportion of patients/caregiver/physician receiving discharge summary | 48 hours post-discharge questionnaire and family physician follow-up phone call
  Proportion of patients/caregiver/physician receiving discharge summary
3-Clinical-level process outcome - Proportion of medication list reconciliation | monthly Chart audit for 4 years
  Proportion of medication list reconciliation
4-Clinical-level process outcome - Proportion of patients with physician appointment | Family physician follow-up phone call post-discharge up to 30 days
  Proportion of patients with physician appointment
5-Clinical-level process outcome - Proportion of patients using telemonitoring | monthly Chart audit for 4 years
  Proportion of patients using telemonitoring using Télé-Surveillance Santé Chaudieres-Appalaches (TSS-CA) database

CONTACTS AND LOCATIONS:
Overall Officials: Patrick M Archambault, MD, MSc, Principal Investigator — Laval University
Locations (1):
- Centres intégrés de santé et de services sociaux (CISSS) De Chaudières-Appalaches, Lévis, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sinha SK, Oakes SL, Chaudhry S, Suh TT. How to Use the ACE Unit to Improve Hospital Safety and Quality for Older Patients: From ACE Units to Elder-Friendly Hospitals. Acute Care for Elders. 2014. pp. 131-156. doi:10.1007/978-1-4939-1025-0_8
- [Background] Sirois MJ, Emond M, Ouellet MC, Perry J, Daoust R, Morin J, Dionne C, Camden S, Moore L, Allain-Boule N. Cumulative incidence of functional decline after minor injuries in previously independent older Canadian individuals in the emergency department. J Am Geriatr Soc. 2013 Oct;61(10):1661-8. doi: 10.1111/jgs.12482. PMID 24117285
- [Background] Reid RC, Cummings GE, Cooper SL, Abel SL, Bissell LJ, Estabrooks CA, Rowe BH, Wagg A, Norton PG, Ertel M, Cummings GG. The Older Persons' Transitions in Care (OPTIC) study: pilot testing of the transition tracking tool. BMC Health Serv Res. 2013 Dec 14;13:515. doi: 10.1186/1472-6963-13-515. PMID 24330805
- [Background] Osborn R, Moulds D, Squires D, Doty MM, Anderson C. International survey of older adults finds shortcomings in access, coordination, and patient-centered care. Health Aff (Millwood). 2014 Dec;33(12):2247-55. doi: 10.1377/hlthaff.2014.0947. Epub 2014 Nov 19. PMID 25410260
- [Background] Dubuc N, Dubois MF, Raiche M, Gueye NR, Hebert R. Meeting the home-care needs of disabled older persons living in the community: does integrated services delivery make a difference? BMC Geriatr. 2011 Oct 26;11:67. doi: 10.1186/1471-2318-11-67. PMID 22029878
- [Background] Levesque JF, Pineault R, Hamel M, Roberge D, Kapetanakis C, Simard B, Prud'homme A. Emerging organisational models of primary healthcare and unmet needs for care: insights from a population-based survey in Quebec province. BMC Fam Pract. 2012 Jul 2;13:66. doi: 10.1186/1471-2296-13-66. PMID 22748060
- [Background] van Walraven C, Taljaard M, Bell CM, Etchells E, Stiell IG, Zarnke K, Forster AJ. A prospective cohort study found that provider and information continuity was low after patient discharge from hospital. J Clin Epidemiol. 2010 Sep;63(9):1000-10. doi: 10.1016/j.jclinepi.2010.01.023. PMID 20656194
- [Background] Haggerty JL, Reid RJ, Freeman GK, Starfield BH, Adair CE, McKendry R. Continuity of care: a multidisciplinary review. BMJ. 2003 Nov 22;327(7425):1219-21. doi: 10.1136/bmj.327.7425.1219. PMID 14630762
- [Background] Trahan LM, Spiers JA, Cummings GG. Decisions to Transfer Nursing Home Residents to Emergency Departments: A Scoping Review of Contributing Factors and Staff Perspectives. J Am Med Dir Assoc. 2016 Nov 1;17(11):994-1005. doi: 10.1016/j.jamda.2016.05.012. Epub 2016 Jun 24. PMID 27349625
- [Background] Dhalla IA, O'Brien T, Ko F, Laupacis A. Toward safer transitions: how can we reduce post-discharge adverse events? Healthc Q. 2012;15 Spec No:63-7. doi: 10.12927/hcq.2012.22839. No abstract available. PMID 22874449
- [Background] Forster AJ, Murff HJ, Peterson JF, Gandhi TK, Bates DW. The incidence and severity of adverse events affecting patients after discharge from the hospital. Ann Intern Med. 2003 Feb 4;138(3):161-7. doi: 10.7326/0003-4819-138-3-200302040-00007. PMID 12558354
- [Background] Coleman EA, Smith JD, Frank JC, Eilertsen TB, Thiare JN, Kramer AM. Development and testing of a measure designed to assess the quality of care transitions. Int J Integr Care. 2002;2:e02. doi: 10.5334/ijic.60. Epub 2002 Jun 1. PMID 16896392
- [Background] Harrison A, Verhoef M. Understanding coordination of care from the consumer's perspective in a regional health system. Health Serv Res. 2002 Aug;37(4):1031-54. doi: 10.1034/j.1600-0560.2002.64.x. PMID 12236382
- [Background] Weaver FM, Perloff L, Waters T. Patients' and caregivers' transition from hospital to home: needs and recommendations. Home Health Care Serv Q. 1998;17(3):27-48. doi: 10.1300/j027v17n03_03. PMID 10351068
- [Background] Beers MH, Sliwkowski J, Brooks J. Compliance with medication orders among the elderly after hospital discharge. Hosp Formul. 1992 Jul;27(7):720-4. PMID 10119187
- [Background] Dudas V, Bookwalter T, Kerr KM, Pantilat SZ. The impact of follow-up telephone calls to patients after hospitalization. Am J Med. 2001 Dec 21;111(9B):26S-30S. doi: 10.1016/s0002-9343(01)00966-4. PMID 11790365
- [Background] van Walraven C, Seth R, Austin PC, Laupacis A. Effect of discharge summary availability during post-discharge visits on hospital readmission. J Gen Intern Med. 2002 Mar;17(3):186-92. doi: 10.1046/j.1525-1497.2002.10741.x. PMID 11929504
- [Background] Moore C, Wisnivesky J, Williams S, McGinn T. Medical errors related to discontinuity of care from an inpatient to an outpatient setting. J Gen Intern Med. 2003 Aug;18(8):646-51. doi: 10.1046/j.1525-1497.2003.20722.x. PMID 12911647
- [Background] Stall N, Nowaczynski M, Sinha SK. Back to the future: home-based primary care for older homebound Canadians: part 1: where we are now. Can Fam Physician. 2013 Mar;59(3):237-40. No abstract available. PMID 23486788
- [Background] Stall N, Nowaczynski M, Sinha SK. Back to the future: home-based primary care for older homebound Canadians: part 2: where we are going. Can Fam Physician. 2013 Mar;59(3):243-5. No abstract available. PMID 23486789
- [Background] Gruneir A, Dhalla IA, van Walraven C, Fischer HD, Camacho X, Rochon PA, Anderson GM. Unplanned readmissions after hospital discharge among patients identified as being at high risk for readmission using a validated predictive algorithm. Open Med. 2011;5(2):e104-11. Epub 2011 May 31. PMID 21915234
- [Background] Jencks SF, Williams MV, Coleman EA. Rehospitalizations among patients in the Medicare fee-for-service program. N Engl J Med. 2009 Apr 2;360(14):1418-28. doi: 10.1056/NEJMsa0803563. PMID 19339721
- [Background] Gill TM, Allore HG, Gahbauer EA, Murphy TE. Change in disability after hospitalization or restricted activity in older persons. JAMA. 2010 Nov 3;304(17):1919-28. doi: 10.1001/jama.2010.1568. PMID 21045098
- [Background] Krumholz HM. Post-hospital syndrome--an acquired, transient condition of generalized risk. N Engl J Med. 2013 Jan 10;368(2):100-2. doi: 10.1056/NEJMp1212324. No abstract available. PMID 23301730
- [Background] Boyd CM, Landefeld CS, Counsell SR, Palmer RM, Fortinsky RH, Kresevic D, Burant C, Covinsky KE. Recovery of activities of daily living in older adults after hospitalization for acute medical illness. J Am Geriatr Soc. 2008 Dec;56(12):2171-9. doi: 10.1111/j.1532-5415.2008.02023.x. PMID 19093915
- [Background] Gill TM, Allore HG, Holford TR, Guo Z. Hospitalization, restricted activity, and the development of disability among older persons. JAMA. 2004 Nov 3;292(17):2115-24. doi: 10.1001/jama.292.17.2115. PMID 15523072
- [Background] Gill TM, Williams CS, Tinetti ME. The combined effects of baseline vulnerability and acute hospital events on the development of functional dependence among community-living older persons. J Gerontol A Biol Sci Med Sci. 1999 Jul;54(7):M377-83. doi: 10.1093/gerona/54.7.m377. PMID 10462171
- [Background] Sirois MJ, Griffith L, Perry J, Daoust R, Veillette N, Lee J, Pelletier M, Wilding L, Emond M. Measuring Frailty Can Help Emergency Departments Identify Independent Seniors at Risk of Functional Decline After Minor Injuries. J Gerontol A Biol Sci Med Sci. 2017 Jan;72(1):68-74. doi: 10.1093/gerona/glv152. Epub 2015 Sep 22. PMID 26400735
- [Background] Covinsky KE, Palmer RM, Fortinsky RH, Counsell SR, Stewart AL, Kresevic D, Burant CJ, Landefeld CS. Loss of independence in activities of daily living in older adults hospitalized with medical illnesses: increased vulnerability with age. J Am Geriatr Soc. 2003 Apr;51(4):451-8. doi: 10.1046/j.1532-5415.2003.51152.x. PMID 12657063
- [Background] Goncalves-Bradley DC, Lannin NA, Clemson LM, Cameron ID, Shepperd S. Discharge planning from hospital. Cochrane Database Syst Rev. 2016 Jan 27;2016(1):CD000313. doi: 10.1002/14651858.CD000313.pub5. PMID 26816297
- [Background] Leppin AL, Gionfriddo MR, Kessler M, Brito JP, Mair FS, Gallacher K, Wang Z, Erwin PJ, Sylvester T, Boehmer K, Ting HH, Murad MH, Shippee ND, Montori VM. Preventing 30-day hospital readmissions: a systematic review and meta-analysis of randomized trials. JAMA Intern Med. 2014 Jul;174(7):1095-107. doi: 10.1001/jamainternmed.2014.1608. PMID 24820131
- [Background] Charles L, Bremault-Phillips S, Parmar J, Johnson M, Sacrey LA. Understanding How to Support Family Caregivers of Seniors with Complex Needs. Can Geriatr J. 2017 Jun 30;20(2):75-84. doi: 10.5770/cgj.20.252. eCollection 2017 Jun. PMID 28690707
- [Background] Ahmed NN, Pearce SE. Acute care for the elderly: a literature review. Popul Health Manag. 2010 Aug;13(4):219-25. doi: 10.1089/pop.2009.0058. PMID 20735247
- [Background] Fox MT, Persaud M, Maimets I, O'Brien K, Brooks D, Tregunno D, Schraa E. Effectiveness of acute geriatric unit care using acute care for elders components: a systematic review and meta-analysis. J Am Geriatr Soc. 2012 Dec;60(12):2237-45. doi: 10.1111/jgs.12028. Epub 2012 Nov 23. PMID 23176020
- [Background] Shepperd S, Iliffe S, Doll HA, Clarke MJ, Kalra L, Wilson AD, Goncalves-Bradley DC. Admission avoidance hospital at home. Cochrane Database Syst Rev. 2016 Sep 1;9(9):CD007491. doi: 10.1002/14651858.CD007491.pub2. PMID 27583824
- [Background] Shepperd S, McClaran J, Phillips CO, Lannin NA, Clemson LM, McCluskey A, Cameron ID, Barras SL. Discharge planning from hospital to home. Cochrane Database Syst Rev. 2010 Jan 20;(1):CD000313. doi: 10.1002/14651858.CD000313.pub3. PMID 20091507
- [Background] Early Supported Discharge Trialists. Services for reducing duration of hospital care for acute stroke patients. Cochrane Database Syst Rev. 2005 Apr 18;(2):CD000443. doi: 10.1002/14651858.CD000443.pub2. PMID 15846604
- [Background] Inglis SC, Clark RA, Dierckx R, Prieto-Merino D, Cleland JG. Structured telephone support or non-invasive telemonitoring for patients with heart failure. Cochrane Database Syst Rev. 2015 Oct 31;2015(10):CD007228. doi: 10.1002/14651858.CD007228.pub3. PMID 26517969
- [Background] McClure R, Turner C, Peel N, Spinks A, Eakin E, Hughes K. Population-based interventions for the prevention of fall-related injuries in older people. Cochrane Database Syst Rev. 2005 Jan 25;2005(1):CD004441. doi: 10.1002/14651858.CD004441.pub2. PMID 15674948
- [Background] Young J, Green J, Forster A, Small N, Lowson K, Bogle S, George J, Heseltine D, Jayasuriya T, Rowe J. Postacute care for older people in community hospitals: a multicenter randomized, controlled trial. J Am Geriatr Soc. 2007 Dec;55(12):1995-2002. doi: 10.1111/j.1532-5415.2007.01456.x. Epub 2007 Nov 2. PMID 17979957
- [Background] Nikolaus T, Specht-Leible N, Bach M, Oster P, Schlierf G. A randomized trial of comprehensive geriatric assessment and home intervention in the care of hospitalized patients. Age Ageing. 1999 Oct;28(6):543-50. doi: 10.1093/ageing/28.6.543. PMID 10604506
- [Background] Green J, Young J, Forster A, Mallinder K, Bogle S, Lowson K, Small N. Effects of locality based community hospital care on independence in older people needing rehabilitation: randomised controlled trial. BMJ. 2005 Aug 6;331(7512):317-22. doi: 10.1136/bmj.38498.387569.8F. Epub 2005 Jul 1. PMID 15994660
- [Background] Coleman EA, Parry C, Chalmers S, Min SJ. The care transitions intervention: results of a randomized controlled trial. Arch Intern Med. 2006 Sep 25;166(17):1822-8. doi: 10.1001/archinte.166.17.1822. PMID 17000937
- [Background] Malone ML, Vollbrecht M, Stephenson J, Burke L, Pagel P, Goodwin JS. AcuteCare for Elders (ACE) tracker and e-Geriatrician: methods to disseminate ACE concepts to hospitals with no geriatricians on staff. J Am Geriatr Soc. 2010 Jan;58(1):161-7. doi: 10.1111/j.1532-5415.2009.02624.x. PMID 20122048
- [Background] Gagliardi AR, Brouwers MC, Bhattacharyya OK. The development of guideline implementation tools: a qualitative study. CMAJ Open. 2015 Jan 13;3(1):E127-33. doi: 10.9778/cmajo.20140064. eCollection 2015 Jan-Mar. PMID 25844365
- [Background] Greenhalgh T, Howick J, Maskrey N; Evidence Based Medicine Renaissance Group. Evidence based medicine: a movement in crisis? BMJ. 2014 Jun 13;348:g3725. doi: 10.1136/bmj.g3725. PMID 24927763
- [Background] McKillop A, Crisp J, Walsh K. Practice guidelines need to address the 'how' and the 'what' of implementation. Prim Health Care Res Dev. 2012 Jan;13(1):48-59. doi: 10.1017/S1463423611000405. Epub 2011 Oct 13. PMID 22008308
- [Background] Dobbins M, Hanna SE, Ciliska D, Manske S, Cameron R, Mercer SL, O'Mara L, DeCorby K, Robeson P. A randomized controlled trial evaluating the impact of knowledge translation and exchange strategies. Implement Sci. 2009 Sep 23;4:61. doi: 10.1186/1748-5908-4-61. PMID 19775439
- [Background] Shekelle PG, Kravitz RL, Beart J, Marger M, Wang M, Lee M. Are nonspecific practice guidelines potentially harmful? A randomized comparison of the effect of nonspecific versus specific guidelines on physician decision making. Health Serv Res. 2000 Mar;34(7):1429-48. PMID 10737446
- [Background] Grilli R, Lomas J. Evaluating the message: the relationship between compliance rate and the subject of a practice guideline. Med Care. 1994 Mar;32(3):202-13. doi: 10.1097/00005650-199403000-00002. PMID 8145598
- [Background] Gagliardi AR, Alhabib S; members of Guidelines International Network Implementation Working Group. Trends in guideline implementation: a scoping systematic review. Implement Sci. 2015 Apr 21;10:54. doi: 10.1186/s13012-015-0247-8. PMID 25895908
- [Background] Pitzul KB, Lane NE, Voruganti T, Khan AI, Innis J, Wodchis WP, Baker GR. Role of context in care transition interventions for medically complex older adults: a realist synthesis protocol. BMJ Open. 2015 Nov 19;5(11):e008686. doi: 10.1136/bmjopen-2015-008686. PMID 26586323
- [Background] Couturier Y, Belzile L, Gagnon D. Principes méthodologiques de l'implantation du modèle PRISMA portant sur l'intégration des services pour les personnes âgées en perte d'autonomie. Management & Avenir. 2011;47: 133
- [Background] Archambault PM, Turgeon AF, Witteman HO, Lauzier F, Moore L, Lamontagne F, Horsley T, Gagnon MP, Droit A, Weiss M, Tremblay S, Lachaine J, Le Sage N, Emond M, Berthelot S, Plaisance A, Lapointe J, Razek T, van de Belt TH, Brand K, Berube M, Clement J, Grajales Iii FJ, Eysenbach G, Kuziemsky C, Friedman D, Lang E, Muscedere J, Rizoli S, Roberts DJ, Scales DC, Sinuff T, Stelfox HT, Gagnon I, Chabot C, Grenier R, Legare F; Canadian Critical Care Trials Group. Implementation and Evaluation of a Wiki Involving Multiple Stakeholders Including Patients in the Promotion of Best Practices in Trauma Care: The WikiTrauma Interrupted Time Series Protocol. JMIR Res Protoc. 2015 Feb 19;4(1):e21. doi: 10.2196/resprot.4024. PMID 25699546
- [Background] Archambault PM, van de Belt TH, Grajales FJ 3rd, Faber MJ, Kuziemsky CE, Gagnon S, Bilodeau A, Rioux S, Nelen WL, Gagnon MP, Turgeon AF, Aubin K, Gold I, Poitras J, Eysenbach G, Kremer JA, Legare F. Wikis and collaborative writing applications in health care: a scoping review. J Med Internet Res. 2013 Oct 8;15(10):e210. doi: 10.2196/jmir.2787. PMID 24103318
- [Background] Archambault PM, Beaupre P, Begin L, Dupuis A, Cote M, Legare F. Impact of Implementing a Wiki to Develop Structured Electronic Order Sets on Physicians' Intention to Use Wiki-Based Order Sets. JMIR Med Inform. 2016 May 17;4(2):e18. doi: 10.2196/medinform.4852. PMID 27189046
- [Background] Archambault PM, Bilodeau A, Gagnon MP, Aubin K, Lavoie A, Lapointe J, Poitras J, Croteau S, Pham-Dinh M, Legare F. Health care professionals' beliefs about using wiki-based reminders to promote best practices in trauma care. J Med Internet Res. 2012 Apr 19;14(2):e49. doi: 10.2196/jmir.1983. PMID 22515985
- [Background] Maher L, Gustafson DH, Evans A. NHS sustainability model. NHS institute for innovation and improvement; 2010
- [Background] Plaisance A, Witteman HO, Heyland DK, Ebell MH, Dupuis A, Lavoie-Berard CA, Legare F, Archambault PM. Development of a Decision Aid for Cardiopulmonary Resuscitation Involving Intensive Care Unit Patients' and Health Professionals' Participation Using User-Centered Design and a Wiki Platform for Rapid Prototyping: A Research Protocol. JMIR Res Protoc. 2016 Feb 11;5(1):e24. doi: 10.2196/resprot.5107. PMID 26869137
- [Background] Cloutier C, Denis JL, Langley A, Lamothe L. Agency at the Managerial Interface: Public Sector Reform as Institutional Work. Journal of Public Administration Research and Theory. 2015;26: 259-276.
- [Background] Anatchkova MD, Barysauskas CM, Kinney RL, Kiefe CI, Ash AS, Lombardini L, Allison JJ. Psychometric evaluation of the Care Transition Measure in TRACE-CORE: do we need a better measure? J Am Heart Assoc. 2014 Jun 4;3(3):e001053. doi: 10.1161/JAHA.114.001053. PMID 24901109
- [Background] Champagne A, Landreville P, Gosselin P, Carmichael PH. Psychometric properties of the French Canadian version of the Geriatric Anxiety Inventory. Aging Ment Health. 2018 Jan;22(1):40-45. doi: 10.1080/13607863.2016.1226767. Epub 2016 Sep 22. PMID 27656951
- [Background] Act P. Revised Statutes of Nova Scotia. Chapter. 1989;208
- [Background] Fleet R, Pelletier C, Marcoux J, Maltais-Giguere J, Archambault P, Audette LD, Plant J, Begin F, Tounkara FK, Poitras J. Differences in access to services in rural emergency departments of Quebec and Ontario. PLoS One. 2015 Apr 15;10(4):e0123746. doi: 10.1371/journal.pone.0123746. eCollection 2015. PMID 25874948
- [Background] Du Plessis V, Beshiri R, Bollman RD, Clemenson H. Definitions of rural. Rural and Small Town Canada Analysis Bulletin. 2001; 3: 1-17
- [Background] Bergman H, Arcand M, Bureau C, Chertkow H, Ducharme F, Joanette Y, et al. Relever le défi de la maladie d'Alzheimer et des maladies apparentées. Une vision centrée sur l'humanisme, la personne et l'excellence. Rapport du comité d'experts en vue de l'élaboration d'un plan national pour la maladie d'Alzheimer. MSSS, gouvernement du Québec; 2009
- [Background] Mosquera I, Vergara I, Larranaga I, Machon M, del Rio M, Calderon C. Measuring the impact of informal elderly caregiving: a systematic review of tools. Qual Life Res. 2016 May;25(5):1059-92. doi: 10.1007/s11136-015-1159-4. Epub 2015 Oct 16. PMID 26475138
- [Background] Mello JA, Macq J, Van Durme T, Ces S, Spruytte N, Van Audenhove C, Declercq A. The determinants of informal caregivers' burden in the care of frail older persons: a dynamic and role-related perspective. Aging Ment Health. 2017 Aug;21(8):838-843. doi: 10.1080/13607863.2016.1168360. Epub 2016 Apr 7. PMID 27054404
- [Background] Penfold RB, Zhang F. Use of interrupted time series analysis in evaluating health care quality improvements. Acad Pediatr. 2013 Nov-Dec;13(6 Suppl):S38-44. doi: 10.1016/j.acap.2013.08.002. PMID 24268083
- [Background] Grimshaw JM, Presseau J, Tetroe J, Eccles MP, Francis JJ, Godin G, Graham ID, Hux JE, Johnston M, Legare F, Lemyre L, Robinson N, Zwarenstein M. Looking inside the black box: results of a theory-based process evaluation exploring the results of a randomized controlled trial of printed educational messages to increase primary care physicians' diabetic retinopathy referrals [Trial registration number ISRCTN72772651]. Implement Sci. 2014 Aug 6;9:86. doi: 10.1186/1748-5908-9-86. PMID 25098442
- [Background] Hsieh HF, Shannon SE. Three approaches to qualitative content analysis. Qual Health Res. 2005 Nov;15(9):1277-88. doi: 10.1177/1049732305276687. PMID 16204405
- [Background] Graham K, Logan J. Using the Ottawa Model of Research Use to implement a skin care program. J Nurs Care Qual. 2004 Jan-Mar;19(1):18-24; quiz 25-6. doi: 10.1097/00001786-200401000-00006. PMID 14717144
- [Background] Leape LL, Berwick DM. Five years after To Err Is Human: what have we learned? JAMA. 2005 May 18;293(19):2384-90. doi: 10.1001/jama.293.19.2384. PMID 15900009
- [Background] Pronovost P, Sexton B, Thompson D. Five years after To Err Is Human. J Crit Care. 2005;20: 76-78
- [Background] Brennan TA, Gawande A, Thomas E, Studdert D. Accidental deaths, saved lives, and improved quality. N Engl J Med. 2005 Sep 29;353(13):1405-9. doi: 10.1056/NEJMsb051157. No abstract available. PMID 16192489
- [Background] Pronovost P, Needham D, Berenholtz S, Sinopoli D, Chu H, Cosgrove S, Sexton B, Hyzy R, Welsh R, Roth G, Bander J, Kepros J, Goeschel C. An intervention to decrease catheter-related bloodstream infections in the ICU. N Engl J Med. 2006 Dec 28;355(26):2725-32. doi: 10.1056/NEJMoa061115. PMID 17192537
- [Background] Middleton S, Lydtin A, Comerford D, Cadilhac DA, McElduff P, Dale S, Hill K, Longworth M, Ward J, Cheung NW, D'Este C; QASCIP Working Group and Steering Committee. From QASC to QASCIP: successful Australian translational scale-up and spread of a proven intervention in acute stroke using a prospective pre-test/post-test study design. BMJ Open. 2016 May 6;6(5):e011568. doi: 10.1136/bmjopen-2016-011568. PMID 27154485
- [Background] Del Mar CB, Green AC, Battistutta D. Do public media campaigns designed to increase skin cancer awareness result in increased skin excision rates? Aust N Z J Public Health. 1997 Dec;21(7):751-4. PMID 9489194
- [Background] Clarke JA, Adams JE. The application of clinical guidelines for skull radiography in the Accident and Emergency department: theory and practice. Clin Radiol. 1990 Mar;41(3):152-5. doi: 10.1016/s0009-9260(05)80957-2. PMID 2323160
- [Background] Ramsay CR, Matowe L, Grilli R, Grimshaw JM, Thomas RE. Interrupted time series designs in health technology assessment: lessons from two systematic reviews of behavior change strategies. Int J Technol Assess Health Care. 2003 Fall;19(4):613-23. doi: 10.1017/s0266462303000576. PMID 15095767
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M. Developing and evaluating complex interventions: the new Medical Research Council guidance. Int J Nurs Stud. 2013 May;50(5):587-92. doi: 10.1016/j.ijnurstu.2012.09.010. Epub 2012 Nov 15. No abstract available. PMID 23159157
- [Background] Hamilton S, McLaren S, Mulhall A. Assessing organisational readiness for change: use of diagnostic analysis prior to the implementation of a multidisciplinary assessment for acute stroke care. Implement Sci. 2007 Jul 14;2:21. doi: 10.1186/1748-5908-2-21. PMID 17629929
- [Background] Grol R, Grimshaw J. Evidence-based implementation of evidence-based medicine. Jt Comm J Qual Improv. 1999 Oct;25(10):503-13. doi: 10.1016/s1070-3241(16)30464-3. PMID 10522231
- [Background] Flodgren G, Parmelli E, Doumit G, Gattellari M, O'Brien MA, Grimshaw J, Eccles MP. Local opinion leaders: effects on professional practice and health care outcomes. Cochrane Database Syst Rev. 2011 Aug 10;(8):CD000125. doi: 10.1002/14651858.CD000125.pub4. PMID 21833939
- [Derived] Archambault PM, Rivard J, Smith PY, Sinha S, Morin M, LeBlanc A, Couturier Y, Pelletier I, Ghandour EK, Legare F, Denis JL, Melady D, Pare D, Chouinard J, Kroon C, Huot-Lavoie M, Bert L, Witteman HO, Brousseau AA, Dallaire C, Sirois MJ, Emond M, Fleet R, Chandavong S; Network Of Canadian Emergency Researchers. Learning Integrated Health System to Mobilize Context-Adapted Knowledge With a Wiki Platform to Improve the Transitions of Frail Seniors From Hospitals and Emergency Departments to the Community (LEARNING WISDOM): Protocol for a Mixed-Methods Implementation Study. JMIR Res Protoc. 2020 Aug 5;9(8):e17363. doi: 10.2196/17363. PMID 32755891
- See also: The Daily - Canada's population estimates: Age and sex, July 1, 2015 [Internet]. 29 Sep 2015 [cited 5 Oct 2016]. — http://www.statcan.gc.ca/daily-quotidien/150929/dq150929b-eng.htm
- See also: Committee on the Learning Health Care System in America, Institute of Medicine. Best Care at Lower Cost: The Path to Continuously Learning Health Care in America [Internet]. — https://market.android.com/details?id=book-_wUw6XCFqGwC
- See also: Cummings GG E al. Older Persons' Transitions in Care (OPTIC): a study protocol. - PubMed - NCBI [Internet]. [cited 19 Oct 2016] — https://www.ncbi.nlm.nih.gov/pubmed/23241360
- See also: Neiterman E E al. Experiences of older adults in transition from hospital to community. - PubMed - NCBI [Internet]. [cited 19 Oct 2016] — https://www.ncbi.nlm.nih.gov/pubmed/25547021
- See also: Mount Sinai first in Canada to Achieve Magnet® Recognition for Nursing Excellence and Patient Care - Mount Sinai Hospital - Toronto [Internet]. [cited 16 Oct 2016] — http://www.mountsinai.on.ca/about_us/news/2015-news/mount-sinai-first-in-canada-to-achieve-magnet-recognition-for-nursing-excellence-and-patient-care
- See also: Knowledge Translation in Health Care: Moving from Evidence to Practice - CIHR [Internet]. 8 Sep 2010 [cited 15 Oct 2016] — http://www.cihr-irsc.gc.ca/e/40618.html
- See also: Projet de loi n°10 : Loi modifiant l'organisation et la gouvernance du réseau de la santé et des services sociaux notamment par l'abolition des agences régionales - Assemblée nationale du Québec [Internet]. [cited 15 Oct 2016] — http://www.assnat.qc.ca/fr/travaux-parlementaires/projets-loi/projet-loi-10-41-1.html
- See also: WikiTrauma [Internet]. [cited 13 Oct 2016] — https://sites.google.com/site/wikitraumaca
- See also: Site internet TSSCA [Internet]. [cited 17 Oct 2016] — http://www.tssca.ca
- See also: Hébert R, Bravo G, Préville M. Reliability, validity and reference values of the Zarit Burden Interview for assessing informal caregivers of community-dwelling older persons with dementia. Canadian Journal on Aging/La Revue canadienne du vieillissement. — https://www.cambridge.org/core/journals/canadian-journal-on-aging-la-revue-canadienne-du-vieillissement/article/reliability-validity-and-reference-values-of-the-zarit-burden-interview-for-assessing-informal-caregivers-of-communitydwelling-older-persons-with-dementia/8D9A9409A5A319B6AAA6B5FD8F54C04D
- See also: Website [Internet]. [cited 16 Oct 2016] — http://www.cihr-irsc.gc.ca/e/40618.html
- See also: [No title] [Internet]. [cited 17 Oct 2016] — http://www.albertahealthservices.ca/org/ahs-org-report-on-structure.pdf
- See also: LEAN QUALITY IMPROVEMENT INITIATIVES | News and Media | Government of Saskatchewan. In: Government of Saskatchewan [Internet]. [cited 17 Oct 2016] — http://www.saskatchewan.ca/government/news-and-media/2011/march/22/lean-quality-improvement-initiatives
- See also: Grol R, Wensing M, Eccles M, Davis D. Improving Patient Care: The Implementation of Change in Health Care [Internet]. Wiley-Blackwell; 2013 — http://books.google.ca/books/about/Improving_Patient_Care.html?hl=&id=K88YYAAACAAJ